CLINICAL TRIAL: NCT06509568
Title: Comparison of Neoadjuvant Chemoradiotherapy Followed by Immunotherapy With Neoadjuvant Chemoimmunotherapy in the Treatment for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma: A Multi-center, Phase II Randomized Clinical Study
Brief Title: Neoadjuvant ChemoRadiotherapy Followed by Immunotherapy and Surgery for Resectable Esophageal Squamous Cell Carcinoma（CRIS-2 Trial）
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang Yang, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-238
Record Dates: First submitted 2024-07-12; First posted 2024-07-19 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant chemoradiotherapy followed by immunotherapy (nCRIT) (Experimental): Patients in the nCRIT group will receive neoadjuvant concurrent chemoradiotherapy: radiation therapy will be administered using IMRT or VMAT with involved-field irradiation at a dose of PTV 41.4 Gy/23 fractions/31 days. Chemotherapy will consist of weekly administration of paclitaxel (albumin-bound) 50 mg/m² and carboplatin (AUC 2) for five weeks, given on the days of radiotherapy. Patients who do not progress on CT and meet immunotherapy criteria will receive fixed-dose tislelizumab (200 mg IV) on days 8 and 29 after chemoradiotherapy, followed by minimally invasive esophagectomy four weeks after completing immunotherapy.
  Interventions: Radiation: Neoadjuvant chemoradiotherapy followed by immunotherapy
- Neoadjuvant chemoimmunotherapy (nCIT) (Active Comparator): Patients in the nCIT group will receive two cycles of TC chemotherapy combined with immunotherapy, specifically paclitaxel (albumin-bound) 100 mg/m² on days 1, 8, 15 or 260mg/m² d1, carboplatin (AUC=5) on days 1, and tislelizumab (200 mg) on days 1. Minimally invasive esophagectomy will be performed 4-6 weeks after completing chemotherapy, and adjuvant immunotherapy is recommended for one year after surgery.
  Interventions: Drug: Neoadjuvant chemoimmunotherapy

INTERVENTIONS:
Radiation: Neoadjuvant chemoradiotherapy followed by immunotherapy — Patients in the nCRIT group will receive neoadjuvant concurrent chemoradiotherapy: radiation therapy will be administered using IMRT or VMAT with involved-field irradiation at a dose of PTV 41.4 Gy/23 fractions/31 days. Chemotherapy will consist of weekly administration of paclitaxel (albumin-bound) 50 mg/m² and carboplatin (AUC 2) for five weeks, given on the days of radiotherapy. Patients who do not progress on CT and meet immunotherapy criteria will receive fixed-dose tislelizumab (200 mg IV) on days 8 and 29 after chemoradiotherapy, followed by minimally invasive esophagectomy four weeks after completing immunotherapy.
  Arms: Neoadjuvant chemoradiotherapy followed by immunotherapy (nCRIT)
Drug: Neoadjuvant chemoimmunotherapy — Patients in the nCIT group will receive two cycles of TC chemotherapy combined with immunotherapy, specifically paclitaxel (albumin-bound) 100 mg/m² on days 1, 8, 15 or 260mg/m² d1, carboplatin (AUC=5) on days 1, and tislelizumab (200 mg) on days 1. Minimally invasive esophagectomy will be performed 4-6 weeks after completing chemotherapy, and adjuvant immunotherapy is recommended for one year after surgery.
  Arms: Neoadjuvant chemoimmunotherapy (nCIT)

SUMMARY:
Based on our previous single-arm Phase Ib study (CRIS trial, NCT06303583), we observed that neoadjuvant chemoradiotherapy followed by immunotherapy (nCRIT) significantly increased the pathological complete response (pCR) rate, achieving approximately 60% in locally advanced esophageal squamous cell carcinoma(ESCC). We plan to initiate a multicenter, prospective, randomized phase II trial designed to compare the efficacy and safety of neoadjuvant chemoimmunotherapy (nCIT) versus neoadjuvant chemoradiotherapy followed by immunotherapy (nCRIT) in treating esophageal squamous cell carcinoma. The primary study population includes patients with operable or potentially operable thoracic ESCC classified as cT3-4aN0 or T2-4aN+ based on endoscopy, enhanced chest and abdominal CT, and whole-body PET scans. Eligible participants are aged 18-75 years with an ECOG performance status of 0-1. Qualified patients will be randomly assigned in a 1:1 ratio to either the nCRIT group or the nCIT group.

Patients in the nCRIT group will receive neoadjuvant concurrent chemoradiotherapy: radiation therapy will be administered using IMRT or VMAT with involved-field irradiation at a dose of PTV 41.4 Gy/23 fractions/31 days. Chemotherapy will consist of weekly administration of paclitaxel (albumin-bound) 50 mg/m² and carboplatin (AUC=2) for five weeks, given on the days of radiotherapy. Patients who do not progress on CT and meet immunotherapy criteria will receive fixed-dose tislelizumab (200 mg IV) on days 8 and 29 after chemoradiotherapy, followed by minimally invasive esophagectomy four weeks after completing immunotherapy.

Patients in the nCIT group will receive two cycles of TC chemotherapy combined with immunotherapy, specifically paclitaxel (albumin-bound) 100 mg/m² on days 1, 8, 15 or 260mg/m² d1, carboplatin (AUC=5) on days 1, and tislelizumab (200 mg) on days 1. Minimally invasive esophagectomy will be performed 4-6 weeks after completing chemotherapy, and adjuvant immunotherapy is recommended for one year after surgery.

The primary endpoint of the study is the pathological complete response (pCR). Secondary endpoints include treatment safety, CT imaging response rate, R0 resection rate, major pathological response (MPR), 2-year event-free survival (EFS), 2-year overall survival (OS) in the intention-to-treat (ITT) population, and analysis of treatment failure reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Age and Consent: Subjects must be male or female, aged ≥18 and ≤75 years at the time of signing the informed consent form.
2. Performance Status: Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1, or a Karnofsky Performance Status (KPS) score of ≥80.
3. Histological Confirmation: Histologically confirmed thoracic esophageal squamous cell carcinoma (ESCC), with the upper boundary of the lesion not exceeding the thoracic inlet.
4. Resectability: Subjects must have resectable or potentially resectable T3-4aN0 or T2-4aN+ ESCC, as per the AJCC/UICC 8th edition clinical staging (cTNM).
5. Lesion Length: The length of the esophageal lesion must be <8 cm.
6. Surgical Eligibility: Subjects must have no contraindications for surgical procedures.
7. Organ Function: Subjects must have good cardiopulmonary function and other organ functions to tolerate chemoradiotherapy and surgery.

   a. Hematology (without the use of any blood components and cell growth factor support treatment within 7 days before the start of study treatment): i. Absolute neutrophil count (ANC) ≥ 1.5×10^9/L (1500/mm^3). ii. Platelet count ≥ 100×10^9/L (100000/mm^3). iii. Hemoglobin ≥ 90 g/L. b. Renal Function: i. Calculated creatinine clearance* (CrCl) ≥ 50 mL/min.

   *CrCl will be calculated using the Cockcroft-Gault formula: CrCl (mL/min) = (140 - age) × weight (kg) × F / (SCr (mg/dL) × 72), where F = 1 for males and 0.85 for females; SCr = serum creatinine. ii. Urine protein < 2+ or 24-hour urine protein quantification < 1.0 g. c. Liver Function: i. Serum total bilirubin (TBiL) ≤ 1.5 × ULN (Upper Limit of Normal). ii. AST and ALT ≤ 2.5 × ULN; for subjects with liver metastasis, AST and ALT ≤ 5 × ULN.

   iii. Serum albumin (ALB) ≥ 28 g/L. d. Coagulation Function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (unless the subject is receiving anticoagulant therapy and INR and APTT are within the expected therapeutic range).

   e. Cardiac Function: Left ventricular ejection fraction (LVEF) ≥ 60%.
8. Female Subjects of Childbearing Potential: Must have a negative urine or serum pregnancy test within 3 days prior to the first dose (if the urine pregnancy test is inconclusive, a serum pregnancy test will be required, and the serum result will be definitive). If a female subject of childbearing potential engages in sexual activity with an unsterilized male partner, she must use highly effective contraception from the start of screening and agree to continue using it for 120 days after the last dose of the study drug. Decisions regarding contraception discontinuation after this period should be discussed with the investigator.
9. Male Subjects with Female Partners of Childbearing Potential: Must use effective contraception from the start of screening until 120 days after the last dose of the study drug. Decisions regarding contraception discontinuation after this period should be discussed with the investigator.
10. Compliance: Subjects must be adequately informed and sign the informed consent form. They must also be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study requirements.

Exclusion Criteria:

1. Cervical esophageal cancer (lesion located in the cervical esophagus).
2. Metastasis to cervical lymph nodes or lymph nodes around the celiac artery.
3. Invasion of the trachea or aorta.
4. Hoarseness caused by the esophageal tumor.
5. Esophageal fistula or a tendency to develop an esophageal fistula.
6. Pregnant or lactating patients.
7. Severe, poorly controlled diabetes mellitus.
8. Inability to use the stomach for esophageal replacement due to previous surgeries.
9. Previous receipt of chemoradiotherapy.
10. Allergy or contraindication to taxane drugs.
11. Inability to provide informed consent due to psychological, familial, or social reasons.
12. History of malignancies other than esophageal cancer.
13. Inability to tolerate chemoradiotherapy due to severe cardiac, pulmonary, hepatic, renal dysfunction, hematologic diseases, or cachexia; BMI < 18.5.
14. Active autoimmune disease, history of autoimmune disease (including but not limited to colitis, hepatitis, hyperthyroidism, etc.), history of immune deficiency (including positive HIV test), or other congenital or acquired immune deficiency disorders, organ transplantation, or allogeneic bone marrow transplantation.
15. Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10^4 copies/mL), active hepatitis C (positive hepatitis C antibody with HCV-RNA levels above the detection limit).
16. History of immunodeficiency; positive HIV antibody test; currently on long-term systemic corticosteroids or other immunosuppressants.
17. Severe infections within 4 weeks prior to the first dose, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; active infections requiring systemic anti-infective therapy within 2 weeks before the first dose (excluding antiviral treatment for hepatitis B or C).
18. Known active tuberculosis (TB); suspected active TB should be ruled out by clinical examination; known active syphilis infection.
19. Receipt of live or attenuated live vaccines within 30 days prior to the first dose or planned receipt of such vaccines during the study period (inactivated vaccines are allowed).
20. History of interstitial lung disease or non-infectious pneumonitis.
21. History of myocarditis, cardiomyopathy, malignant arrhythmias; unstable angina requiring hospitalization, myocardial infarction, congestive heart failure (NYHA class 2 or above), or vascular disease (e.g., aneurysms at risk of rupture) within 12 months prior to the first dose; or other cardiac conditions that may affect the safety evaluation of the study drug (e.g., poorly controlled arrhythmias, myocardial ischemia).
22. Known psychiatric disorders, drug abuse, alcoholism, or a history of substance abuse.
23. Local or systemic diseases caused by non-malignant tumors; or diseases or symptoms secondary to tumors that may lead to high medical risk and/or uncertainty in survival assessment, such as tumor leukemoid reaction (white blood cell count > 20×10^9/L), cachexia (e.g., known weight loss of more than 10% in the 3 months prior to screening).
24. Any condition that the investigator believes may pose a risk to the subject's participation in the study, interfere with the evaluation of the study drug, or affect the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
pCR | 1 months after surgery
  Pathologic complete response (pCR) was defined as the absence of cancer cells in both the esophagus and lymph nodes following neoadjuvant chemoradiotherapy

SECONDARY OUTCOMES:
R0 resection rate | 1 months after surgery
  R0 resection rate refers to the proportion of patients who undergo a surgical procedure to remove a tumor and achieve a complete resection with no residual microscopic disease.
MPR | 1 months after surgery
  Major pathological response (MPR) is a measure of neoadjuvant immunotherapy efficacy. It is defined as having no more than 10% residual viable tumor cells by routine hematoxylin and eosin (H&E) staining after therapy.
2-year EFS | 2 years after randomization
  Event-Free Survival (EFS) refers to the length of time after the treatment starts during which a patient remains free from certain negative events, such as disease progression, recurrence, or death from any cause.
2-year OS | 2 years after randomization
  Time from randomization to any death
Adverse Events | 2 years after randomization
  any undesirable experiences or side effects that occur in a patient during the trial
HRQoL | 2 years after randomization
  Health-Related Quality of Life (HRQoL) refers to a patient's overall well-being, encompassing physical, mental, and social aspects of health as they are affected by a medical condition or its treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Izutsu M, Kobayashi S, Higuchi N, Yuasa Y, Ogawa K, Narimatsu Y, Nakano K, Hiramatsu K, Shen Y, Azemoto S. [CT angiography of the liver]. Nihon Igaku Hoshasen Gakkai Zasshi. 1993 Jan 25;53(1):101-3. Japanese. PMID 8441593
- [Background] Qin J, Xue L, Hao A, Guo X, Jiang T, Ni Y, Liu S, Chen Y, Jiang H, Zhang C, Kang M, Lin J, Li H, Li C, Tian H, Li L, Fu J, Zhang Y, Ma J, Wang X, Fu M, Yang H, Yang Z, Han Y, Chen L, Tan L, Dai T, Liao Y, Zhang W, Li B, Chen Q, Guo S, Qi Y, Wei L, Li Z, Tian Z, Kang X, Zhang R, Li Y, Wang Z, Chen X, Hou Z, Zheng R, Zhu W, He J, Li Y. Neoadjuvant chemotherapy with or without camrelizumab in resectable esophageal squamous cell carcinoma: the randomized phase 3 ESCORT-NEO/NCCES01 trial. Nat Med. 2024 Sep;30(9):2549-2557. doi: 10.1038/s41591-024-03064-w. Epub 2024 Jul 2. PMID 38956195